CLINICAL TRIAL: NCT00963287
Title: Trial of Chinese Prescription on Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHTCM-003
Record Dates: First submitted 2009-06-11; First posted 2009-08-21 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2009-08

CONDITIONS: Ulcerative Colitis
Keywords: alternative medicine; traditional Chinese medicine
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bascial prescription (Experimental): Decoction ,two times a day,one bag of decoction one time
  Interventions: Drug: bascial prescription plus or minus herbs depend on symptoms
- low does of bascial decoction (Placebo Comparator): Decoction ,two times a day, one bag decoction of one time
  Interventions: Drug: bascial prescription plus or minus herbs depend on symptoms

INTERVENTIONS:
Drug: bascial prescription plus or minus herbs depend on symptoms — Decoction ,two times a day

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the Chinese prescription on Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ulcerative colitis
* Male of female patients between 18-65 years old
* Written informed consent

Exclusion Criteria:

* Combine with malignant pathology on epithelial dysplasia of mucosa
* Combined with severe heart, gallbladder, kidney, endocrine system, hemopoietic system or nervous system disease.
* Pregnancy or breast feeding women, or unwilling to have contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Histopathological examination,enteroscopy,blood test,symptoms ,pulse tracings,tongue demonstration | 8 weeks

SECONDARY OUTCOMES:
Indicates of liver and renal function | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xie Jianqun, Phd, Study Director — Shanghai University of Chinese Medicine
Locations (1):
- Longhua hospital, Shanghai, Shanghai Municipality, China